CLINICAL TRIAL: NCT04862572
Title: Investigating Disinhibitory Brain Mechanism in Tinnitus and Hearing Loss: Is There a Maladaptive Signature of Auditory Cortex GABA Loss and Dysconnectivity?
Brief Title: Investigating Disinhibitory Brain Mechanism in Tinnitus and Hearing Loss
Acronym: IGNITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 21020
Record Dates: First submitted 2021-03-22; First posted 2021-04-28 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Tinnitus; Hearing Loss
Keywords: Tinnitus; Hearing loss; Inhibition; Functional connectivity; Structural connectivity
MeSH Terms: conditions — Tinnitus; Hearing Loss; Inhibition, Psychological

STUDY DESIGN:
Intervention Model Description: Cross sectional case-control multimodal MRI, audio- and psychometric study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- People with tinnitus (Experimental): People with tinnitus will undergo all interventions (audiology test, MRI scans, tinnitus-related questionnaires).
  Interventions: Other: MRI scanning
- People without tinnitus (Experimental): People with tinnitus will undergo most of all interventions (audiology test, MRI scans) except filling up the tinnitus-related questionnaires.
  Interventions: Other: MRI scanning

INTERVENTIONS:
Other: MRI scanning — In the audiological assessment, participants will undergo various audiometric test, such as pure tone audiometry with extended high-frequency range, speech audiometry, tympanometry, and auditory reflex threshold. These tests are all noninvasive and aim to assess participants hearing threshold, speech-in-noise difficulty, whether or not they have conductive hearing loss, and test efferent auditory function. The appointment will take around 60-90 minutes. An experienced audiologist on-site will be in charge of this procedure.
  In the MRI appointment, participant will undergo MRI scanning. Before the MRI scan, a researcher with experienced radiographer will re-check that the participant is safe to be scanned, with the standard University of Nottingham safety questionnaire. This rechecking step is necessary to make sure that participants are still eligible for the scanning. An experience radiographer will be in charge of this procedure.
  Other Names: Audiological assessment

SUMMARY:
Tinnitus, the perception of sound in the absence of an external acoustic stimulus. Tinnitus is often perceived inside the head rather than the ear and is a common condition with a prevalence estimated between 10 and 15% in adults. Between 1 and 3% of this population are having a significant impact on their quality of life. Despite its high prevalence, the underlying mechanisms of tinnitus still remain unclear.

The majority of tinnitus cases associated with some degree of hearing loss, making hearing loss the biggest risk factor for tinnitus. Recently, it has been suggested that hearing deficits, such as speech-in-noise difficulty, can exist in the absence of any overt hearing loss within the audiometric range (0.125-8 kHz). This is referred to as "hidden hearing loss" and has been suggested to be associated with hearing loss at above-audiometric (> 8 kHz) frequencies.

This project is aimed at studying the underlying mechanisms of tinnitus and the possible relation with overt or hidden hearing loss. Specifically, the investigators want to test the hypothesis that tinnitus is caused by maladaptive plasticity arising as a result of auditory input deprivation. This idea is supported by the finding that tinnitus may disappear when the hearing, and thus auditory input, recover. Disruptions at lower levels of the auditory pathway could lead to alterations in synaptic transmission and neurotransmitter release in more central regions of the auditory system (e.g., in the auditory cortex). This may create an imbalance between neuronal excitation and inhibition, and re-routing of auditory pathways, leading to abnormal neural excitability and connectivity.

In this study, the investigators question whether auditory cortex disinhibition is specifically related to tinnitus, or is a consequence of hearing loss. To answer this question, the investigators propose to conduct a study that aims to investigate the inhibition mechanism by quantifying GABA concentration level, neural activity and functional connectivity strength of auditory cortex using non-invasive imaging techniques, namely Magnetic Resonance Spectroscopy (MRS) and functional Magnetic Resonance Imaging (fMRI). The investigators expected to possibly provide a tinnitus biomarker, and this may help to direct future treatments.

DETAILED DESCRIPTION:
SELECTION AND WITHDRAWAL OF PARTICIPANTS

Recruitment

1. Clinical routes Suitable candidates may be identified by the sites, at Ropewalk House Nottingham Audiology Services and ear, nose, and throat (ENT) services at Nottingham University Hospitals National Health Service (NHS) trust, via searches of their clinical databases or opportunistically during routine clinical appointments. Candidates will only be approached by a member of staff at the site or NIHR Clinical Research Network (CRN) staff to whom recruitment activities have been delegated by the local PI. All patient contact information will be kept confidential and undisclosed to the research team. The initial approach will be providing the participant with the information packs, that will contain (i) an invitation letter, (ii) a participant information sheet explaining all aspects pertaining to participation in the study and (iii) a reply slip. Potential participants who wish to find out more about the study will then be able to opt to be contacted by the researcher by completing a reply slip attached to the invitation letter and returning it in a pre-paid and addressed envelope. Alternatively, potential participants can contact the researcher directly via email and phone number that is written on the participant information sheet.

   It will be explained to the potential participant that entry into the trial is entirely voluntary and that their treatment and care will not be affected by their decision. It will also be explained that they can withdraw at any time, but attempts will be made to avoid this occurrence. In the event of their withdrawal, it will be explained that their data collected so far cannot be erased and the investigators will seek consent to use the data in the final analyses where appropriate.

   Posters about the study will be on display in the relevant clinical areas.
2. Non-clinical routes:

   Non-clinical routes will include advertising the study via
   * Invitation emails to NIHR Nottingham Hearing participant database. This database includes everyone that previously stating interest to takes part in tinnitus and hearing loss study (including healthy participants and hearing-related patients).
   * Newsletter articles and announcements published by the relevant patient and professional organisations.
   * Posts on social media channels (Twitter (@hearingnhir, @TIN_ACT @UoNPIBeacon) and Facebook.

   In all cases, fully informed consent will be sought by explaining the study's procedures and requirements following the standard script to interested potential participants. The potential participants will have ideally a minimum of 24 hours in which to decide whether or not to take part in this study. If the participant agrees to take part in the study, the consent form will be signed, during COVID-19 time this will be done electronically. In all cases, informed consent will be obtained and the consent form will have to be signed prior to any assessment or intervention.

   Expected duration of participant participation

   The study is expected to run between August 2021 until April 2022. The expected total duration of participation in the study from the time of informed consent is likely to range from one week to eight weeks. This prolonged time estimate is due to possible organisational difficulties in arranging the audiology assessment and the MRI scans, especially during the COVID-19 pandemic. There will be two visits for each participant, where each visit will last for around 1.5 hours.

   Removal of participants from therapy or assessments/Participant Withdrawal

   Participants may choose to withdraw from the study at any time without giving a reason. They will be withdrawn from the study if they are unable to be scanned (due to uncontrollable movement), or if they are unable for any reason to complete the audiology assessment. Participants will also be removed in the event of pregnancy, taking GABA enhancing or anti-depressants medication, having a cochlear or any metal implant that is not compatible with MRI scan, or having metal implant(s) during the time that they first agree to participate and the booked date for scanning, or withdrawal of consent.

   In the unique case relating to COVID-19, if participants report symptoms of the virus before the study appointment, it will be discussed if they still want to continue participating in the study, and while waiting for their 14 days quarantine the investigators will reschedule their appointment. However, in the case where participants are confirmed to have coronavirus before the study appointment, participants will be removed from the study.

   Participants will be made aware (via the information sheet and consent form) that should they withdraw the data collected to date cannot be erased and may still be used in the final analysis. If a participant withdraws from the study, the investigators will record the reason for and date of discontinuation. They will be replaced, such that at the end of the study, the number of completed scans, not the number of enrolled participants defines the end. Abrupt termination of enrolment in the study will not affect participant safety. The participants will be made aware that this will not affect their future care.

   STATISTICS

   Methods

   The investigators will use three tests to analyse the data: primary, secondary, and exploratory test.

   + Primary test

   Univariate group comparison between-group differences in imaging outcomes, this includes a comparison between:

   Auditory cortex GABA, GABA/Glx, and Cho level, Auditory cortex cerebral blood flow (CBF), Local functional connectivity density, Interhemispheric auditory cortices functional connectivity, Cross-modal functional connectivity between auditory and visual cortex, and Auditory cortex blood oxygen level-dependent (BOLD) response to visual attention task.

   Between-group test for differences in correlation, between:

   GABA and hearing loss, and Auditory cortex functional connectivity and hearing loss.

   + Secondary test: Within-group correlation analysis of imaging markers of inhibition (such as GABA, functional connectivity, CBF and BOLD response to attention) with audiometric results indexing sensory deafferentation. The investigators will also do regression analysis of imaging metrics with tinnitus severity.

   + Exploratory: Multivariate prediction model of tinnitus severity and regression of brain network metrics with affective tinnitus phenotypes.

   The findings will be evaluated by the investigator team. Due to the complex statistic question and strategy, the investigators will seek advice throughout the analysis from both experienced statistician and senior researcher. The analysis will take place on the University of Nottingham (UoN) computers, using R statistical software package and Matlab, and backed up to the UoN servers.

   Sample size and justification

   Approximately 60 subjects in total (30 per group). For details, please see below. All tests were done using the R statistical software package and STATA SE16.

   GABA

   Previous studies investigating GABA alteration in tinnitus and hearing loss patients are very limited, with the discrepancy between them. In Gao's study with a total sample of 36 subjects, reported around 50% (r=-0.57) of total GABA variance is explained by hearing loss in the elderly cohort, with the assumption that half of their subjects have tinnitus (tin+) and the rest of the half did not have tinnitus (tin-), while in Sedley's study with a total sample of 28 subjects, reported significant GABA concentration reduced (median 1.12 vs 1.28 mM/L) in right auditory cortex for tin+ > tin- respectively.

   Using these values, the investigators can estimate their effect size using:

   Cohen's d = (M_1-M_2)/(SD pooled) Also, Cohen's d = 2r/√(1-r^2 )

   Where effect size for Gao and Sedley's study respectively are, r=-0.57 (correlation between hearing loss and GABA) and d=-3.7 (GABA effect size between patient and control). One might think of this as a promising effect, but the investigators are aware of the low power of these studies considering their small sample size compared to the population, and thus these effect sizes might be inflated and not represent the true effect size.

   The investigators then propose to recruit a bigger sample size, and with the time constraint and the limitation due to the COVID-19 pandemic, the realistic number of subjects that the investigators are pursuing is 30 per group (N total=60). With this sample size and based on knowledge from previous studies, the investigators estimated effect size of d=0.7 (two-sided test) and r=0.4 using 0.05 alpha value and 80% power.

   The investigators will also use a relative measurement to quantify GABA such as GABA/Cr ratio that presumably has a lower variance, and thus will power the effect size, compared to the absolute measure (i.e., mM/L).

   Previous pilot measurement has shown that GABA measurement was good enough in terms of repeatability and showing the right trend but failed to reach significance in within-subject measurement. Therefore, the other strategy is to involve and inter-relate the GABA measurement with other functional measures (resting-, visual task, tonotopy scan). The analysis will not be limited to only between-subject analysis, but the investigators will also do within-subject analysis that has shown to have more robust results.

   Functional connectivity

   In fMRI, the combination of a large number of dependent variables (i.e. huge number of voxel comparison) and a relatively small number of observations (subjects) resulted in underpowered studies with grossly inflated effect size and thus poorly represent the actual effects in the full sample/population. However, using meta-analysis, one can study whether reported findings from selected pooled studies (with a small sample) are really significant or not.

   Similar to the GABA approach, the investigators then estimate the effect size from a meta-analysis study of functional changes between tin + and tin - and compared it with the estimated effect size.

   r = z/√N Cohen's d = 2r/√(1-r^2 )

   The investigators estimate to be able to detect medium effect size, d=0.6 (N total= 30, whole brain, 0.05 alpha value, and 80% power).

   As the investigators are fully aware that the results might not represent the full picture of the true effect, the proposed study will still benefit tinnitus field research and add more power to validate previous findings. It is also noted that the meta-analysis study was using a whole-brain measurement (i.e. ReHo), where high variance is expected due to the big number of voxel comparison.

   Instead, the study proposes to focus on region-of-interest (ROIs) analysis to lower the variance, thus increasing the effect size. Defining the ROIs will be guided by an independent condition such as visual task and tonotopy scan, using Independent Component Analysis (ICA) analysis, and/or using anatomical maps such as Brodmann area. Some functional measures that will be applied are regional connectivity density, interregional correlations, and fractional amplitude of low-frequency fluctuations (fALFF). Cross-validation with GABA measurement, both between-subject and within-subject is expected to enrich the current knowledge between inhibition and neural activation changes in tinnitus patients.

   Procedures for missing, unused and spurious data

   In the case of missing or spurious data, the participants whose data is in question will be excluded from that particular analysis.

ELIGIBILITY:
Inclusion Criteria:

* Are age 18-80 years.
* Are eligible to be scanned using MRI and to undergo audiometry and psychometry.
* Are able to give informed consent.
* Must have a good comprehension of English in order to complete the hearing-related questionnaires

Exclusion Criteria:

* Pregnant women will be excluded based on MRI safety recommendations.
* Past medical history of acoustic neuroma and Ménière's disease.
* Significant past medical history that may affect brain GABA and functional metrics such as stroke, multiple sclerosis, epilepsy, diabetes, cardiovascular, major neurodegenerative or psychiatric conditions, cancer requiring systemic chemotherapy or brain radiotherapy.
* Individuals who had in last 3 months and/or currently taking a sedating or GABA enhancing or psychoactive drugs (opioids, anti-depressants).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
GABA neurotransmitter level measured using MRS and neural activity and connectivity strength in auditory resting-state networks using functional MRI scan. | During 3-6 months after the data has been collected
  Primary test:
  * Univariate group comparison between-group differences in imaging outcomes: auditory cortex GABA, local functional connectivity density (REHO), interhemispheric auditory cortices functional connectivity, cross-modal functional connectivity between auditory and visual cortex, auditory cortex neural activity (using BOLD response) to visual attention task.
  * Between-group test for differences in correlation: GABA and hearing loss, auditory cortex functional connectivity and hearing loss.

SECONDARY OUTCOMES:
Measures of GABA level in the auditory cortex and correlation with tinnitus severity scores and tinnitus negative affect scores. | During 3-6 months after the data has been collected
  Secondary test:
  * Within-group correlation analysis of GABA level with audiometric results indexing sensory deafferentation.
  * Regression analysis of GABA level with tinnitus severity.
Measures of neural activity, and connectivity changes in brain-wide and correlation of these measures with tinnitus severity scores and tinnitus negative affect scores. | During 3-6 months after the data has been collected
  Secondary test:
  * Within-group correlation analysis of functional connectivity and neural activity to attention) with audiometric results indexing sensory deafferentation.
  * Regression analysis of functional connectivity and neural activity with tinnitus severity.

CONTACTS AND LOCATIONS:
Overall Officials: Dorothee Auer, Prof., Study Director — University of Nottingham; Anissa Ramadhani, Principal Investigator — University of Nottingham
Locations (3):
- United Kingdom (3):
  - Greater Nottingham and Midlands areas, Nottingham
  - NIHR Hearing Research, Nottingham
  - Nottingham Audiology clinics, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the University of Nottingham's, the Government's, and our funders' policies the research data may be shared with researchers in other universities and organizations, including those in other countries, for research in health and social care. Data sharing in this way is usually anonymized. Although the detail of what and how to share them will need to be followed up.
Supporting Information: Analytic Code
Time Frame: Data will become available 3 months after the last data acquisition. They will be available up to 3 years.

REFERENCES:
- [Background] Alain C, Roye A, Salloum C. Effects of age-related hearing loss and background noise on neuromagnetic activity from auditory cortex. Front Syst Neurosci. 2014 Jan 31;8:8. doi: 10.3389/fnsys.2014.00008. eCollection 2014. PMID 24550790
- [Background] Auerbach BD, Rodrigues PV, Salvi RJ. Central gain control in tinnitus and hyperacusis. Front Neurol. 2014 Oct 24;5:206. doi: 10.3389/fneur.2014.00206. eCollection 2014. PMID 25386157
- [Background] Baguley D, McFerran D, Hall D. Tinnitus. Lancet. 2013 Nov 9;382(9904):1600-7. doi: 10.1016/S0140-6736(13)60142-7. Epub 2013 Jul 2. PMID 23827090
- [Background] Bauer CA. Tinnitus. N Engl J Med. 2018 Mar 29;378(13):1224-1231. doi: 10.1056/NEJMcp1506631. No abstract available. PMID 29601255
- [Background] Bauer CA, Turner JG, Caspary DM, Myers KS, Brozoski TJ. Tinnitus and inferior colliculus activity in chinchillas related to three distinct patterns of cochlear trauma. J Neurosci Res. 2008 Aug 15;86(11):2564-78. doi: 10.1002/jnr.21699. PMID 18438941
- [Background] Deco G, Ponce-Alvarez A, Hagmann P, Romani GL, Mantini D, Corbetta M. How local excitation-inhibition ratio impacts the whole brain dynamics. J Neurosci. 2014 Jun 4;34(23):7886-98. doi: 10.1523/JNEUROSCI.5068-13.2014. PMID 24899711
- [Background] Demeester K, van Wieringen A, Hendrickx JJ, Topsakal V, Fransen E, Van Laer L, De Ridder D, Van Camp G, Van de Heyning P. Prevalence of tinnitus and audiometric shape. B-ENT. 2007;3 Suppl 7:37-49. PMID 18225607
- [Background] Dempsey MF, Condon B, Hadley DM. MRI safety review. Semin Ultrasound CT MR. 2002 Oct;23(5):392-401. doi: 10.1016/s0887-2171(02)90010-7. PMID 12509109
- [Background] Eggermont JJ, Roberts LE. Tinnitus: animal models and findings in humans. Cell Tissue Res. 2015 Jul;361(1):311-36. doi: 10.1007/s00441-014-1992-8. Epub 2014 Sep 30. PMID 25266340
- [Background] Eggermont JJ, Tass PA. Maladaptive neural synchrony in tinnitus: origin and restoration. Front Neurol. 2015 Feb 17;6:29. doi: 10.3389/fneur.2015.00029. eCollection 2015. PMID 25741316
- [Background] Gao F, Wang G, Ma W, Ren F, Li M, Dong Y, Liu C, Liu B, Bai X, Zhao B, Edden RA. Decreased auditory GABA+ concentrations in presbycusis demonstrated by edited magnetic resonance spectroscopy. Neuroimage. 2015 Feb 1;106:311-6. doi: 10.1016/j.neuroimage.2014.11.023. Epub 2014 Nov 15. PMID 25463460
- [Background] Gao Y, Manzoor N, Kaltenbach JA. Evidence of activity-dependent plasticity in the dorsal cochlear nucleus, in vivo, induced by brief sound exposure. Hear Res. 2016 Nov;341:31-42. doi: 10.1016/j.heares.2016.07.011. Epub 2016 Aug 1. PMID 27490001
- [Background] Hoffman, H. J., & Reed, G. W. (2004). Epidemiology of tinnitus. Tinnitus: Theory and management, 16, 16-41.
- [Background] Ito T, Brincat SL, Siegel M, Mill RD, He BJ, Miller EK, Rotstein HG, Cole MW. Task-evoked activity quenches neural correlations and variability across cortical areas. PLoS Comput Biol. 2020 Aug 3;16(8):e1007983. doi: 10.1371/journal.pcbi.1007983. eCollection 2020 Aug. PMID 32745096
- [Background] Kalappa BI, Brozoski TJ, Turner JG, Caspary DM. Single unit hyperactivity and bursting in the auditory thalamus of awake rats directly correlates with behavioural evidence of tinnitus. J Physiol. 2014 Nov 15;592(22):5065-78. doi: 10.1113/jphysiol.2014.278572. Epub 2014 Sep 12. PMID 25217380
- [Background] Kaltenbach JA, Afman CE. Hyperactivity in the dorsal cochlear nucleus after intense sound exposure and its resemblance to tone-evoked activity: a physiological model for tinnitus. Hear Res. 2000 Feb;140(1-2):165-72. doi: 10.1016/s0378-5955(99)00197-5. PMID 10675644
- [Background] Kim JY, Kim YH, Lee S, Seo JH, Song HJ, Cho JH, Chang Y. Alteration of functional connectivity in tinnitus brain revealed by resting-state fMRI? A pilot study. Int J Audiol. 2012 May;51(5):413-7. doi: 10.3109/14992027.2011.652677. Epub 2012 Jan 30. PMID 22283490
- [Background] C Kohrman D, Wan G, Cassinotti L, Corfas G. Hidden Hearing Loss: A Disorder with Multiple Etiologies and Mechanisms. Cold Spring Harb Perspect Med. 2020 Jan 2;10(1):a035493. doi: 10.1101/cshperspect.a035493. PMID 30617057
- [Background] Kotak VC, Fujisawa S, Lee FA, Karthikeyan O, Aoki C, Sanes DH. Hearing loss raises excitability in the auditory cortex. J Neurosci. 2005 Apr 13;25(15):3908-18. doi: 10.1523/JNEUROSCI.5169-04.2005. PMID 15829643
- [Background] Koush Y, de Graaf RA, Kupers R, Dricot L, Ptito M, Behar KL, Rothman DL, Hyder F. Metabolic underpinnings of activated and deactivated cortical areas in human brain. J Cereb Blood Flow Metab. 2021 May;41(5):986-1000. doi: 10.1177/0271678X21989186. Epub 2021 Jan 20. PMID 33472521
- [Background] Lefeuvre J, Chedeau J, Boulet M, Fain G, Papon JF, Nguyen Y, Nevoux J. Hidden hearing loss and tinnitus: Utility of the high-definition audiograms in diagnosis. Clin Otolaryngol. 2019 Nov;44(6):1170-1175. doi: 10.1111/coa.13435. Epub 2019 Oct 4. No abstract available. PMID 31535428
- [Background] Lockwood AH, Salvi RJ, Burkard RF. Tinnitus. N Engl J Med. 2002 Sep 19;347(12):904-10. doi: 10.1056/NEJMra013395. No abstract available. PMID 12239260
- [Background] Middleton JW, Kiritani T, Pedersen C, Turner JG, Shepherd GM, Tzounopoulos T. Mice with behavioral evidence of tinnitus exhibit dorsal cochlear nucleus hyperactivity because of decreased GABAergic inhibition. Proc Natl Acad Sci U S A. 2011 May 3;108(18):7601-6. doi: 10.1073/pnas.1100223108. Epub 2011 Apr 18. PMID 21502491
- [Background] Moller AR. The role of neural plasticity in tinnitus. Prog Brain Res. 2007;166:37-45. doi: 10.1016/S0079-6123(07)66003-8. PMID 17956769
- [Background] Nondahl DM, Cruickshanks KJ, Wiley TL, Klein R, Klein BE, Tweed TS. Prevalence and 5-year incidence of tinnitus among older adults: the epidemiology of hearing loss study. J Am Acad Audiol. 2002 Jun;13(6):323-31. PMID 12141389
- [Background] Norena AJ, Farley BJ. Tinnitus-related neural activity: theories of generation, propagation, and centralization. Hear Res. 2013 Jan;295:161-71. doi: 10.1016/j.heares.2012.09.010. Epub 2012 Oct 23. PMID 23088832
- [Background] Roberts LE, Eggermont JJ, Caspary DM, Shore SE, Melcher JR, Kaltenbach JA. Ringing ears: the neuroscience of tinnitus. J Neurosci. 2010 Nov 10;30(45):14972-9. doi: 10.1523/JNEUROSCI.4028-10.2010. PMID 21068300
- [Background] Schaette R, Kempter R. Development of tinnitus-related neuronal hyperactivity through homeostatic plasticity after hearing loss: a computational model. Eur J Neurosci. 2006 Jun;23(11):3124-38. doi: 10.1111/j.1460-9568.2006.04774.x. PMID 16820003
- [Background] Schreiber BE, Agrup C, Haskard DO, Luxon LM. Sudden sensorineural hearing loss. Lancet. 2010 Apr 3;375(9721):1203-11. doi: 10.1016/S0140-6736(09)62071-7. PMID 20362815
- [Background] Sedley W, Parikh J, Edden RA, Tait V, Blamire A, Griffiths TD. Human Auditory Cortex Neurochemistry Reflects the Presence and Severity of Tinnitus. J Neurosci. 2015 Nov 4;35(44):14822-8. doi: 10.1523/JNEUROSCI.2695-15.2015. PMID 26538652
- [Background] Shore SE, Roberts LE, Langguth B. Maladaptive plasticity in tinnitus--triggers, mechanisms and treatment. Nat Rev Neurol. 2016 Mar;12(3):150-60. doi: 10.1038/nrneurol.2016.12. Epub 2016 Feb 12. PMID 26868680
- [Background] Vielsmeier V, Lehner A, Strutz J, Steffens T, Kreuzer PM, Schecklmann M, Landgrebe M, Langguth B, Kleinjung T. The Relevance of the High Frequency Audiometry in Tinnitus Patients with Normal Hearing in Conventional Pure-Tone Audiometry. Biomed Res Int. 2015;2015:302515. doi: 10.1155/2015/302515. Epub 2015 Oct 25. PMID 26583098
- [Background] Xiong B, Liu Z, Liu Q, Peng Y, Wu H, Lin Y, Zhao X, Sun W. Missed hearing loss in tinnitus patients with normal audiograms. Hear Res. 2019 Dec;384:107826. doi: 10.1016/j.heares.2019.107826. Epub 2019 Oct 17. PMID 31683074
- [Background] Yang S, Weiner BD, Zhang LS, Cho SJ, Bao S. Homeostatic plasticity drives tinnitus perception in an animal model. Proc Natl Acad Sci U S A. 2011 Sep 6;108(36):14974-9. doi: 10.1073/pnas.1107998108. Epub 2011 Sep 6. PMID 21896771
- See also: Project website — https://www.tinact.eu/